CLINICAL TRIAL: NCT02603302
Title: Phase II Study of Neoadjuvant Radiotherapy Dose Escalation in Association With Chemotherapy for the Treatment of Locally Advanced Rectal Cancer
Brief Title: Radiation Dose Escalation in Locally Advanced Rectal Cancer
Acronym: RaDE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Marcos Santos, MD PhD, University of Brasilia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; radiotherapy; escalated dose; interval
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Locally advanced rectal cancer (Experimental): RT (3D conformal RT) 45 Gy to the whole pelvis + boost 14.4 Gy to the GTV + Chemotherapy with 5-FU
  Surgery 8 weeks after the neoadjvuant treatment.
  Interventions: Radiation: Dose Escalation Radiotherapy; Procedure: Delayed surgery

INTERVENTIONS:
Radiation: Dose Escalation Radiotherapy — RT (3D conformal RT) 45 Gy to the whole pelvis + boost 14.4 Gy to the GTV Chemotherapy with 5-FU
Procedure: Delayed surgery — Surgery after 8 weeks with TME (total mesorectal excision)

SUMMARY:
This is a one arm study where patients with locally advanced rectal cancer will receive neoadjuvant treatment with escalated dose radiotherapy (with 3D conformal radiotherapy, up to 59,4 Gy) and radiosensitizing chemotherapy. Then, patients will operated (total mesorectal excision) after 8 weeks of interval. Primary endpoint will be pCR (pathologic complete response).

DETAILED DESCRIPTION:
Introduction:

Rectal cancer is a highly prevalent disease all over the world. In Brazil, it is the second most common cancer among women (after breast tumors), with an estimated incidence of 17.2 cases per 100,000 inhabitants and is the third most common cancer in men (after prostate and lung cancers), with an estimated incidence of 15.4 cases per 100,000 inhabitants.

Goals:

The aim of this study is to evaluate the pathologic complete response (pCR) of patients with locally advanced rectal cancer (LARC) treated with neoadjuvant radiochemotherapy (RCT) employing anticancer drugs at standard dose and interval extended to surgery with or without adjuvant neoplastic therapy.

Procedures:

Neoadjuvant chemoradiotherapy with radiation dose escalation associated with radiosensitizing therapy and surgery with a total mesorectal excision (TME), 8 weeks after completing neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced rectal cancer, 0-15 cm from anal verge, cT3/4 or cN+

Exclusion Criteria:

* Metastatic disease, previous chemotherapy, previous radiotherapy, previous malignant non-skin tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | Through study completion, an average of 2 years
  Pathologic evaluation of the surgical specimen

SECONDARY OUTCOMES:
Disease free survival | 2 years
  Evaluation of disease free survival
Overall survival | 2 years
  Evaluation of overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Santos, MD PhD, Study Chair — Brasília University
Locations (1):
- Brasilia Univeristy Hospital, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We may share data in requested by metanalists